CLINICAL TRIAL: NCT04067037
Title: Single-arm, Multi-center and Phase II Clinical Trial of Camrelizumab Combined With AVD (Epirubicin, Vincristine and Dacarbazine) in the First-line Treatment for Patients With Advanced Classical Hodgkin's Lymphoma
Brief Title: Camrelizumab Combined With AVD in the First-line Treatment for Patients With Advanced Classical Hodgkin's Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanyan Liu, Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYY01
Record Dates: First submitted 2019-08-18; First posted 2019-08-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Classical Hodgkin Lymphoma; PD-1/PD-L1 Signaling Pathway; Camrelizumab
MeSH Terms: interventions — camrelizumab; Epirubicin; Vincristine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab Combined With AVD regimen (Experimental): Camrelizumab 200mg, Intravenous administration on day 1 and day 15 combined with regimen：AVD (Epirubicin, Vincristine and Dacarbazine): repeated every 4 weeks, up to 6 cycles.
  Interventions: Drug: Camrelizumab; Drug: Epirubicin; Drug: Vincristine; Drug: Dacarbazine

INTERVENTIONS:
Drug: Camrelizumab — 200mg, Intravenous administration on day 1 and day 15 of each 4-week cycle until disease progression or unacceptable toxicity develops, up to 6 cycles.
  Other Names: SHR-1210
Drug: Epirubicin — 35mg/m2, Intravenous administration on day 1 and day 15 of each 4-week cycle until disease progression or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Epirubicin hydrochloride
Drug: Vincristine — 1.4mg/m2, Intravenous administration on day 1 and day 15 of each 4-week cycle until disease progression or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Oncovin
Drug: Dacarbazine — 375mg/m2, Intravenous administration on day 1 and day 15 of each 4-week cycle until disease progression or unacceptable toxicity develops, up to 6 cycles.

SUMMARY:
This is a prospective single-arm, multi-center and phase II clinical trial to observe the efficacy and safety of Camrelizumab combined with AVD in the first-line treatment for patients with advanced classical Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Hodgkin's lymphoma (HL) is a kind of malignant tumor of the lymph system, approximately 95% of which are classical hodgkin's lymphoma (cHL). Currently, ABVD and BEACOPP are commonly used in the first-line treatment for cHL. There are about one third of patients, whose pre-treatment assessment are mainly advanced cHL, suffering relapse and drug resistance. PD-1/PD-L1 signaling pathway plays an important role in the development and progression of cHL. Nivolumab and Pembrolizumab have been used in the therapy in relapsed and refractory patients with cHL. Camrelizumab, a humanized anti-PD-1 IgG4 monoclonal antibody, is independently developed in China. The goal of our trial is to assess the efficacy and safety of Camrelizumab combined with AVD (Epirubicin, Vincristine and Dacarbazine) in the first-line treatment for patients with advanced classical Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years old (including 18 and 75)
2. Diagnosed as advanced classical hodgkin's lymphoma based on histopathology
3. Subjects must be untreated (Ann Arbor Stage III/IV or Ann Arbor II with B symptoms along with mediastinal big tumor or extranodal changes)
4. No receiving chemotherapy before enrollment
5. Having at least one measurable lesions
6. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-2
7. Life expectancy no less than 3 months
8. enough main organ function
9. Pregnancy test within 7 days must be negative for women of childbearing period, and appropriate measures should be taken for contraception for women in childbearing period during the study and six months after this study
10. Agreeing to sign the written informed consents

Exclusion Criteria:

1. Diagnosed as nodular lymphocyte predominant lymphoma or grey-zone lymphoma
2. Diagnosed as central nervous system lymphoma
3. usage of immunosuppressants before enrollment and the dose of immunosuppressant used >10mg / day oral prednisone for more than 2 weeks
4. Previously treated with anti-PD-1/PD-L1/PD-L2/CTLA-4
5. Active autoimmune disease
6. Vaccination with anti-tumor vaccine or other immune treatments less than 3 months
7. Serious surgery and trauma less than two weeks
8. Other malignant tumor history or active malignant tumor need be treated
9. Systemic therapy for serious acute/chronic infection
10. Congestive heart failure, uncontrolled coronary heart disease, arrhythmia and heart infarction less than 6 months
11. Active tuberculosis
12. Vaccination with live attenuated vaccine less than 4 weeks
13. HIV-positive, AIDS patients and untreated active hepatitis
14. Researchers determine unsuited to participate in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
complete metabolic response rate (CMRR) | every 8 weeks from the day of the first cycle of treatment to 4 weeks after the completion of 6 cycles of treatment after the last patient's enrollment (each cycle is 28 days)
  the proportion of patients who achieved a complete metabolic response (CMR) as their best overall response (BOR) from the first dose of study treatment through the end-of-treatment (EOT) assessment

SECONDARY OUTCOMES:
objective response rate | every 8 weeks from the day of the first cycle of treatment to 4 weeks after the completion of 6 cycles of treatment after the last patient's enrollment (each cycle is 28 days)
  the total proportion of patients with complete response (CR) and partial response (PR)
duration of complete response(DoCR) | The time from the date of first documented complete response until the date of first documented disease recurrence, progression, or death from any cause, whichever occurs first, assessed up to 10 years.
  The time from the date of first documented complete response until the date of first documented disease recurrence, progression, or death from any cause, whichever occurs first.
2-year progression-free survival | from the day of the first cycle of treatment to the date of confirmed progressive disease or death, whichever occurs first, up to 2 years after last patient's enrollment (each cycle is 28 days)
  the total proportion of patients with no progression from date of the first day of treatment to the date of confirmed progressive disease or death which one occurrs first
overall survival | from date of the first cycle of treatment to the date of death from any cause, assessed up to 10 years (each cycle is 28 days)
  from date of first day of treatment to the date of death by any cause
incidence and relationship with study drugs of grade 3-4 adverse events and abnormal laboratory examinations | from the date of the first cycle of treatment to 1 year after last patient's enrollment (each cycle is 28 days)
  the incidence and relationship with study drugs of grade 3 or 4 adverse events (based on NCI CTC-AE v4.03) and abnormal laboratory examinations

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Liu, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (3):
- China (3):
  - An Yang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital, and College of Clinical Medicine of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan